CLINICAL TRIAL: NCT04477876
Title: Study of CD160, an Activating NK Cell Receptor, in Melanoma: a Potential Therapeutic Target?
Acronym: NKCD160MEL
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190953
Record Dates: First submitted 2020-05-11; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although immunotherapy revolutionized melanoma outcomes over the last 10 years, only 40-50% of patients respond to treatments and 25% develop acquired resistances. Natural Killer (NK) cells naturally recognize and kill tumor cells. However, the immunosuppressive micro-environment generated by the tumor decreases NK cells' killing activity. CD160 is a NK cell receptor identified and characterized in our laboratory. Engagement of the GPI isoform (CD160-GPI) initiates NK cell cytotoxic response. Upon NK cell activation, a transmembrane isoform (CD160-TM) is neo-synthesized which promotes the amplification of activated NK cell cytotoxicity.

The aim of this study is to assess the phenotypic profile of advanced stages melanoma patients' NK cells (mainly CD160-TM expression or its induction) and therefore the therapeutic potential of the use of an anti-CD160-TM agonist antibody to boost the NK-dependent mechanism leading to tumor depletion.

ELIGIBILITY:
Inclusion Criteria :

* Patients aged18-years old or over
* ECOG score between 0-2
* Inoperable stage III or stage IV melanoma
* Naïve of treatment or in progression after one or several treatment lines
* Give their written consent for the present study and be included in MelBase cohort.
* health insurance coverage.

Supplementary inclusion criteria for part II :

* skin or subcutaneous melanoma lesions
* agree and inform consent for a cutaneous biopsy or a tumor sample if presenting lymph nodes involvement if part of the usual clinical practice.

Exclusion Criteria:

* Pregnant and breastfeeding women
* Patients with psychiatric disorders
* Patients already included in another clinical trial
* Having received chemotherapy or radiotherapy during the last 4 weeks,
* Patient presenting another solid or blood cancer, chronic viral infection (e.g. HIV, HBV or HCV)
* Been treated with more than 10mg of steroids until the 4 weeks before inclusion.
* Refusal to participate to the study
* Patients under guardianship or curatorship
* Patients on state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inoperable stage III/ stage IV melanoma patients
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of effector cells activation and degranulation (CD69 and CD107a staining ) | at inclusion
  Difference between cells incubated with the anti CD160-TM antibody and with isotipic control ab ( flow cytometry)

SECONDARY OUTCOMES:
Overall survival | at 1 year post inclusion
Overall survival | at 2 years post inclusion
Overall survival | at 3 years post inclusion
Overall survival | at 4 years post inclusion
Overall survival | at 5 years post inclusion
Progression free survival | at 1 year
Progression free survival | at 2 years
Progression free survival | at 3 years
Progression free survival | at 4 years
Progression free survival | at 5 years
Objective response rate | at one year
Objective response rate | at 2 years
Objective response rate | at 3 years
Objective response rate | at 4 years
Objective response rate | at 5 years
Phenotypic characteristics of NK cells | at inclusion
  Assessment by flow cytometry of the expression levels of activating or inhibitory receptors (e.g. CD160-GPI, NKp46), phenotypic markers (e.g CD16, CD3), as well as activation (CD69) and degranulation (CD107a) markers by the NK cell population (defined as CD3- CD56+ cell). Results will be expressed as the % of positive cells for each marker among the NK cell population
cytokine profile | at inclusion
  Assessment by flow cytometry using a cytokine beads array (BD Biosciences) of the Th1/Th2/Th17 cytokine content. The presence of the following cytokine will be assessed: IL17-A, IFN-g, TNF, IL10, IL-6, IL-4 and IL-2. The mean fluorescence intensities will be recorded and quantifications will be done, using an individual standard curve, for each cytokine. Results will be expressed in pg/ml.
Détection and quantification of sCD160 in patients' serum | at inclusion

IPD SHARING:
Plan to Share IPD: Undecided